CLINICAL TRIAL: NCT05183971
Title: Early Detection of Proprioceptive Dysfunction in Degenerative Cervical Myelopathy by Proprioceptive Functional Analysis in Activities of Daily Living
Brief Title: Proprioceptive Deficits in Degenerative Cervical Myelopathy
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 20-746
Record Dates: First submitted 2021-12-14; First posted 2022-01-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Cervical Myelopathy
Keywords: Degenerative Cervical Myelopathy; Proprioceptive Deficits

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- (1) Degenerative Cervical Myelopathy: Chinese subjects aged 50 or above who have radiological evidence of Degenerative Cervical Myelopathy, symptomatic with Nurick Grade less than 3 will be included.
  Interventions: Other: Proprioceptive Functional Analysis System
- (2) Healthy Controls: Chinese healthy controls aged 50 or above who have no myelopathic signs of Degenerative Cervical Myelopathy with Nurick Grade less than 3 will be included.
  Interventions: Other: Proprioceptive Functional Analysis System

INTERVENTIONS:
Other: Proprioceptive Functional Analysis System — Proprioceptive testing and Physical Performance Tests

SUMMARY:
Proprioceptive deficits in degenerative cervical myelopathy (DCM) is a progressive neurological deficits in somatosensory and motor function which affects the body balance and motor control. DCM usually presents with body incoordination, hand clumsiness and gait disturbance associated with proprioceptive dysfunction that hinders the physical performance and functions. In this study, a non-invasive assessment protocol on proprioception will be developed for detecting subtle proprioceptive deficits at the early stage of disease through simple Physical Performance Tests for population older than 45. By adopting the physical performance tests as the diagnostic predictors of DCM, we aim to avoid the development of devastating consequences and disabilities.

DETAILED DESCRIPTION:
DCM is a chronic insidious disease, one of the most disabling orthopaedic conditions, which involves compression of the spinal cord by the surrounding structures in cervical spinal region. It characterizes with progressive neurological deficits in body coordination, hand clumsiness and gait disturbance as the preliminary symptom which may cause by proprioceptive dysfunction .

Physical performance and function hinder patients' hand clumsiness, gait disturbance and body imbalance. The incoordination between body, upper limbs and lower limbs will be resulted from proprioceptive deficits caused by spinal cord compression. By adopting the Proprioceptive Functional Analysis System (PFAS), proprioceptive deficits over the core body joints and peripheral joints could be tested during Activity of Daily Living (ADL) with reference to normal subjects' performance. All subjects will be tested by the PFAS and Physical Performance Tests.

The idea of regional proprioceptive deficit will be incorporated in the assessment protocol for DCM to facilitates a breakthrough from the traditional DCM functional evaluation.

In developing a non-invasive assessment protocol to assess proprioceptive deficit, we aim to detect subtle proprioceptive deficit from the tests, especially at the very early stage of disease. We target to demonstrate the validity of Physical Performance Tests are evenly high as that of the advanced technology, PFAS.

Consequently, by adopting the valid Physical Performance Tests in health screening scheme for population older than 45 within the community can serve as an early diagnostic parameter of DCM and avoid delayed treatment leading to devastating consequences and disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* Aged 50 or above
* With radiological evidence of degenerative cervical myelopathy, both symptomatic and asymptomatic
* Nurick grade less than 3

Exclusion Criteria:

* Non-Chinese ethnicity
* Aged under 50
* without any radiological proof of cervical myelopathy
* Active problems of tuberculosis spine, lumbar spinal diseases, and other problems causing pain or deformities over the limbs that may affect their balance and movement
* Presents with extra-pyramidal or other disorders involving the cerebellum or frontal lobe of the cerebrum leading to poor balance and gait disturbance
* Previous spinal operation with residual disturbance in balance or gait
* Non-communicable patients with insufficient cognitive ability to express their symptoms clearly
* Non-walker
* Blind or deaf

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Radiologically confirmed with Degenerative Cervical Myelopathy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2035-09-30 (Estimated); Study Completion 2036-09-30 (Estimated)

PRIMARY OUTCOMES:
Modified Japanese Orthopaedics Association Scoring System for Cervical Myelopathy (mJOA) | 15 years
  mJOA is a self-reported functional questionnaire on disease severity through assessing 4 domains:
  1. Upper Limb Function
  2. Lower Limb Function
  3. Sensory Function
  4. Bladder Function
  mJOA has a total score of 17 and it categories DCM patient into different severity as below:
  1. Mild >= 15
  2. Moderate = 12-14
  3. Severe < 12

SECONDARY OUTCOMES:
Proprioceptive Deficits - Speed Test | 15 years
  Proprioceptive deficits hinder the limb coordination, especially the fine finger dexterity, reciprocal walking and stepping. Thus, incoordination over the lower and upper limbs will then be resulted and which alters the speed and integrity of the performance in the Physical Performance Tests validated for DCM.
  In the physical performance tests, it has divided into 2 separate sections, the "Speed Test" will be recorded for in terms of the "Time required to complete" the standardized test process in seconds
Proprioceptive Deficits - Time Limited Test | 15 years
  Time Limited Test of physical performance test will be assessed and data will be recorded in terms of "Total number of repetitions completed" within strictly fixed time frame

CONTACTS AND LOCATIONS:
Overall Officials: Karlen Ka Pui Law, M. Phil, Principal Investigator — The University of Hong Kong
Locations (1):
- The Duchess of Kent Children's Hospital at Sandy Bay, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Data should not be shared with other researchers